CLINICAL TRIAL: NCT03138785
Title: UVX as an Adjuvant in the Treatment of Fungal Keratitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Farabi Eye Hospital (Other)
Responsible Party: Principal Investigator, mohammad soleimani, assistant professor, Farabi Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32768
Record Dates: First submitted 2017-02-22; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Treatment
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment (Experimental): In this arm, patients with documented fungal keratitis undergo conventional medical treatment.
  Interventions: Drug: topical voriconazole / levofloxacin systemic itraconazole
- conventional treatment +CXL (Active Comparator): In this arm, patients with documented fungal keratitis undergo conventional medical treatment plus CXL, beginning on the first day
  Interventions: Drug: topical voriconazole / levofloxacin systemic itraconazole; Radiation: CXL

INTERVENTIONS:
Drug: topical voriconazole / levofloxacin systemic itraconazole — starting topical voriconazole every hour tapering after 4 days , levofloxacin every 6 hours, Itraconazole 100mg /BD for 2 weeks
Radiation: CXL — 30 min Riboflavin prescription to the cornea followed by 30 min UV-A radiation at 3mW/cm2 associated with Riboflavin administration
  Other Names: Collagen cross-linking/ UVx
  Arms: conventional treatment +CXL

SUMMARY:
In this study, investigators want to find the effect of adjuvant collagen cross-linking in the treatment of fungal keratitis

ELIGIBILITY:
Inclusion Criteria:

* fungal keratitis documented by culture or confocal scanning without any previous treatment

Exclusion Criteria:

* Previous treatment
* Thinning at presentation
* Perforation
* Associated with other microbial or viral keratitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-01 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
time of complete healing (days) | 180 days
  time to scar formation (days)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558